CLINICAL TRIAL: NCT04978727
Title: A Pilot Study of Safety, Tolerability, and Immunological Effects of SurVaxM in Pediatric Patients With Progressive or Relapsed Medulloblastoma, High Grade Glioma, Ependymoma and Newly Diagnosed Diffuse Intrinsic Pontine Glioma
Brief Title: A Pilot Study of SurVaxM in Children Progressive or Relapsed Medulloblastoma, High Grade Glioma, Ependymoma and Newly Diagnosed Diffuse Intrinsic Pontine Glioma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: Roswell Park Cancer Institute (Other); National Cancer Institute (NCI) (NIH); American Lebanese Syrian Associated Charities (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBTC 060; UM1CA081457 (NIH); NCI-2021-07694 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-060 (Other: Pediatric Brain Tumor Consortium); PBTC-060 (Other: CTEP)
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Medulloblastoma; Glioblastoma Multiforme; Anaplastic Astrocytoma; High-grade Astrocytoma NOS; Anaplastic Oligodendroglioma; Anaplastic Ependymoma; Ependymoma; Diffuse Intrinsic Pontine Glioma
Keywords: SurVaxM
MeSH Terms: conditions — Medulloblastoma; Glioblastoma; Astrocytoma; Oligodendroglioma; Ependymoma; Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention/treatment in disease specific or age stratified fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- SurVaxM for patients with relapsed or progressive MB, HGG or ependymoma ages ≥10 and ≤21 years (Experimental): 500 mcg (1 mL) SurVaxM emulsion with Montanide ISA 51. Sargramostim dose is 3.33 mcg/kg/dose for patients < 30 kg, and 100 mcg for patients ≥ 30 kg.
  Priming Phase: patients will get one dose of SurVaxM combined with Montanide ISA 51 through a subcutaneous injection at the start of the study and every 2 weeks for 6 weeks (for a total of 4 doses). At each SurVaxM/Montanide ISA 51 injection, patients will also get an injection of sargramostim.
  Maintenance Phase: the patient will get a SurVaxM/Montanide ISA 51 dose along with a sargramostim dose about every 8 weeks for up to two years.
  After finishing study treatment, patients will be followed for up to 3 years following the last dose of SurVaxM/Montanide ISA 51. Patients will be followed in clinic every 3 months during the follow-up.
  Interventions: Biological: SurVaxM for patients with relapsed or progressive MB, HGG or ependymoma ages ≥10 and ≤21 years
- SurVaxM for patients with relapsed or progressive MB, HGG or ependymoma ages ≥1 and <10 years (Experimental): 500 mcg (1 mL) SurVaxM emulsion with Montanide ISA 51. Sargramostim dose is 3.33 mcg/kg/dose for patients < 30 kg, and 100 mcg for patients ≥ 30 kg.
  Priming Phase: patients will get one dose of SurVaxM combined with Montanide ISA 51 through a subcutaneous injection at the start of the study and every 2 weeks for 6 weeks (for a total of 4 doses). At each SurVaxM/Montanide ISA 51 injection, patients will also get an injection of sargramostim.
  Maintenance Phase: the patient will get a SurVaxM/Montanide ISA 51 dose along with a sargramostim dose about every 8 weeks for up to two years.
  After finishing study treatment, patients will be followed for up to 3 years following the last dose of SurVaxM/Montanide ISA 51. Patients will be followed in clinic every 3 months during the follow-up.
  Interventions: Biological: SurVaxM for patients with relapsed or progressive MB, HGG or ependymoma ages ≥1 and <10 years
- SurVaxM for patients with non-relapsed DIPG post radiation-therapy ages ≥1 and ≤21 years (Experimental): 500 mcg (1 mL) SurVaxM emulsion with Montanide ISA 51. Sargramostim dose is 3.33 mcg/kg/dose for patients < 30 kg, and 100 mcg for patients ≥ 30 kg.
  Priming Phase: patients will get one dose of SurVaxM combined with Montanide ISA 51 through a subcutaneous injection at the start of the study and every 2 weeks for 6 weeks (for a total of 4 doses). At each SurVaxM/Montanide ISA 51 injection, patients will also get an injection of sargramostim.
  Maintenance Phase: the patient will get a SurVaxM/Montanide ISA 51 dose along with a sargramostim dose about every 8 weeks for up to two years.
  After finishing study treatment, patients will be followed for up to 3 years following the last dose of SurVaxM/Montanide ISA 51. Patients will be followed in clinic every 3 months during the follow-up.
  Interventions: Biological: SurVaxM for patients with non-relapsed DIPG post radiation-therapy ages ≥1 and ≤21 years

INTERVENTIONS:
Biological: SurVaxM for patients with relapsed or progressive MB, HGG or ependymoma ages ≥10 and ≤21 years — 500 mcg (1 mL) SurVaxM emulsion with Montanide ISA 51. Sargramostim dose is 3.33 mcg/kg/dose for patients < 30 kg, and 100 mcg for patients ≥ 30 kg.
  Arms: SurVaxM for patients with relapsed or progressive MB, HGG or ependymoma ages ≥10 and ≤21 years
Biological: SurVaxM for patients with relapsed or progressive MB, HGG or ependymoma ages ≥1 and <10 years — 500 mcg (1 mL) SurVaxM emulsion with Montanide ISA 51. Sargramostim dose is 3.33 mcg/kg/dose for patients < 30 kg, and 100 mcg for patients ≥ 30 kg.
  Arms: SurVaxM for patients with relapsed or progressive MB, HGG or ependymoma ages ≥1 and <10 years
Biological: SurVaxM for patients with non-relapsed DIPG post radiation-therapy ages ≥1 and ≤21 years — 500 mcg (1 mL) SurVaxM emulsion with Montanide ISA 51. Sargramostim dose is 3.33 mcg/kg/dose for patients < 30 kg, and 100 mcg for patients ≥ 30 kg.
  Arms: SurVaxM for patients with non-relapsed DIPG post radiation-therapy ages ≥1 and ≤21 years

SUMMARY:
Patients will receive a vaccine called SurVaxM on this study. While vaccines are usually thought of as ways to prevent diseases, vaccines can also be used to treat cancer. SurVaxM is designed to tell the body's immune system to look for tumor cells that express a protein called survivin and destroy them. The survivin protein can be found on up to 95% of glioblastomas and other types of cancer but is not found in normal cells. If the body's immune system knows to destroy cells that express survivin, it may help to control tumor growth and recurrence.

SurVaxM will be mixed with Montanide ISA 51 before it is given. Montanide ISA 51 is an ingredient that helps create a stronger immune response in people, which helps the vaccine work better.

This study has two phases: Priming and Maintenance. During the Priming Phase, patients will get one dose of SurVaxM combined with Montanide ISA 51 through a subcutaneous injection (a shot under the skin) at the start of the study and every 2 weeks for 6 weeks (for a total of 4 doses). At the same time that patients get the SurVaxM/Montanide ISA 51 injection, they will also get a second subcutaneous injection of a medicine called sargramostim. Sargramostim is given close to the SurVaxM//Montanide ISA 51 injection and works to stimulate the immune system to help the SurVaxM/Montanide ISA 51 work more effectively.

If a patient completes the Priming Phase without severe side effects and his or her disease stays the same or improves, he or she can continue to the Maintenance Phase. During the Maintenance Phase, the patient will get a SurVaxM/Montanide ISA 51 dose along with a sargramostim dose about every 8 weeks for up to two years.

After a patient finishes the study treatment, the doctor and study team will continue to follow his/her condition and watch for side effects up to 3 years following the last dose of SurVaxM/Montanide ISA 51. Patients will be seen in clinic every 3 months during the follow-up period.

DETAILED DESCRIPTION:
This is a multicenter pilot study of SurVaxM (SVN53-67/M57-KLH) for children and young adults with progressive or relapsed medulloblastoma, high grade glioma, ependymoma and newly diagnosed diffuse intrinsic pontine glioma.

Survivin (BIRC5) is an inhibitor of apoptosis (IAP) protein that is highly expressed in many cancers. Survivin's high level of expression in certain pediatric malignancies makes it an attractive molecular target for new therapies, including active specific vaccination-based immunotherapy.

The design of the SurVaxM vaccine employs several strategies to create an effective antitumor immunogen, including: 1) incorporation of multiple MHC class I epitopes, 2) peptide modification to enhance binding to certain MHC class I molecules, 3) cytokine helper support, and 4) antibody-mediated tumor cell killing. All of these effects would not be expected with the unmodified class-I restricted short survivin peptides employed in previously studied glioma vaccines.

There are no prior clinical trials of SurVaxM in pediatric patients; however, SurVaxM has been studied in several adult trials, including a phase I study conducted at Roswell Park Comprehensive Cancer Center. Following the single-institution phase I trial, a multicenter phase IIa trial (NCT024455557) was conducted in 63 patients with newly diagnosed glioblastoma. All patients in this study underwent surgical resection of their tumors. Patients then underwent chemoradiation with temozolomide according to the Stupp protocol. This was followed by a one-month hiatus from chemotherapy, during which priming doses of SurVaxM were initiated. The priming phase of vaccination was then followed by initiation of standard adjuvant chemotherapy with temozolomide and maintenance doses of SurVaxM as an add-on to standard chemotherapy. There have been no regimen-limiting toxicities (RLT) or grade ≥ 3 SAE attributable to SurVaxM, with most toxicities being related to temozolomide. The most common AE was grade 1-2 injection site reaction with 2 patients experiencing Montanide-related granulomatous panniculitis with local skin ulceration at vaccine injection sites, both of which resolved. Humoral and survivin-specific CD8+ T cell responses were observed in almost all patients. Twelve-month overall survival (OS12) was 86% from first immunization and 93.4% from diagnosis. OS12 for meMGMT was 93.1% and unMGMT was 78% from first immunization. Median time to tumor progression (mPFS) was 13.9 months from diagnosis. Although not a randomized trial, these results are superior to overall survival reported in various studies in which patients received standard of care treatment for this disease. A randomized phase IIb clinical trial of standard therapy plus SurVaxM is currently being developed with intent for drug registration, if successful.

The primary objective of this trial is to assess the toxicity profile of SurVaxM in emulsion with Montanide plus sargramostim in children with relapsed or progressive medulloblastoma and high-grade glioma, ependymoma and non-recurrent diffuse intrinsic pontine glioma post-radiation therapy. Patients will be enrolled into three separate strata based on age and diagnosis. Enrollment will be staged to allow for safety evaluations between strata.

Each patient will receive 500 micrograms SurVaxM as a 1:1 mixture with Montanide ISA 51 in a water-in-oil emulsion. The SurVaxM-Montanide emulsion injection will be followed immediately by sargramostim (or biosimilar) given via a second separate subcutaneous injection in close proximity to the vaccine injection site. Patients will receive four injections administered over a 6-week period, followed by 14 days of follow-up, called the Priming Phase (8 weeks total). Beginning 8 weeks after the fourth priming dose, a maintenance dose of SurVaxM with Montanide ISA 51 may be given every 8 weeks (± 2 weeks) for two years or until an off-treatment criterion is met.

ELIGIBILITY:
Screening Inclusion Criteria:

* • DIAGNOSIS: Patients with a histologically confirmed diagnosis of a primary CNS tumor that is progressive or recurrent defined as radiographic progression in any known residual tumor, or the appearance of one or more new lesions, leptomeningeal disease, or new cerebrospinal fluid (CSF) positivity for malignant cells, after most recent treatment modality. At the time of diagnosis or recurrence, all tumors must have histologic verification of one of the following:

  * Medulloblastoma
  * Glioblastoma multiforme (GBM)
  * Anaplastic astrocytoma
  * High-grade astrocytoma, NOS
  * Anaplastic oligodendroglioma
  * Anaplastic ependymoma (WHO Grade III)
  * Ependymoma (WHO Grade II)

Diffuse Intrinsic Pontine Gliomas (DIPG) Patients:

Patients with newly diagnosed diffuse intrinsic pontine gliomas (DIPGs), defined as tumors with a pontine epicenter and diffuse involvement of 2/3 or more of the pons, are eligible without histologic confirmation and will proceed directly to enrollment without screening.

• TUMOR TISSUE- Patients must provide tumor tissue (3 unstained slides or paraffin block) to determine their survivin expression status.

Demonstration of survivin expression of at least 1% on tumor tissue by immunohistochemistry is required and must be performed in the central laboratory at Roswell Park Comprehensive Cancer Center (RPCCC) to confirm eligibility.

* Age: Patients must be ≥ 1 year of age and ≤ 21 years of age at the time of screening.
* Screening Consent: Participant is willing to sign a screening consent. The screening consent is to be obtained according to institutional guidelines. Assent, when appropriate, will be obtained according to institutional guidelines.
* Potential Eligibility for Study Enrollment: Patients screened for this trial should be expected to meet the criteria for treatment.

Enrollment Inclusion Criteria:

• DIAGNOSIS: Patients with a histologically confirmed diagnosis of a primary CNS tumor that is progressive or recurrent defined as progression in any known residual tumor, or the appearance of one or more new lesions, or new cerebrospinal fluid (CSF) positivity for malignant cells, after having failed standard therapy. At the time of diagnosis or recurrence, all tumors must have histologic verification of one of the following:

* Medulloblastoma
* Glioblastoma multiforme (GBM)
* Anaplastic astrocytoma
* High-grade astrocytoma, NOS
* Anaplastic oligodendroglioma
* Anaplastic ependymoma (WHO Grade III)
* Ependymoma (WHO Grade II)

Patients with newly diagnosed DIPG: Patients with diffuse intrinsic pontine gliomas (DIPGs) will be eligible 14 to 56 days post-completion of radiation therapy if they do not have any evidence of progression.

* Patients with a typical DIPG on MR imaging, defined as a tumor with a pontine epicenter and diffuse involvement of more than 2/3 of the pons, are eligible without histologic confirmation.

  o Note: Patients with typical DIPG who undergo a biopsy are eligible provided the tumor is a diffuse glioma WHO Grade II-IV with OR without H3 K27M mutation.
* Patients with pontine lesions that do not meet these MR imaging criteria will be eligible if there is histologic confirmation of diffuse glioma WHO Grade II-IV with H3 K27M mutation.
* DEMONSTRATION OF SURVIVIN EXPRESSION: For patients with relapsed or progressive medulloblastoma, HGG, or ependymoma, demonstration of survivin expression as assessed after screening consent/assent of at least 1% on tumor tissue by immunohistochemistry (ICH) is required and must have been performed in the central laboratory at Roswell Park Comprehensive Cancer Center (RPCCC) to confirm eligibility. For patients with DIPG, diagnostic biopsy for histologic confirmation is not required, and tumor expression of survivin is therefore not required for eligibility for these patients.
* DISEASE STATUS: Patients must have evaluable disease within the central nervous system to be eligible. Evaluable disease includes either measurable OR non-measurable disease, defined as follows:

Measurable disease: bi-dimensionally measurable disease; at least one lesion that can be accurately measured in at least two dimensions (per protocol guidelines).

* Non-measurable disease:

  * A lesion that does not meet the criteria for measurable disease as defined above; or
  * diffuse leptomeningeal disease, or
  * no tumor visible on imaging but presence of malignant cells on cytologic examination of CSF.
* AGE:

  * Stratum 1 (progressive or recurrent) patients must be ≥10 years of age and ≤ 21 years of age at the time of study screening.
  * Stratum 2 (progressive or recurrent) patients must be ≥1 year of age and < 10 years of age at the time of study screening.
  * Stratum 3 (newly diagnosed DIPG) patients must be ≥1 year of age and ≤ 21 years of age at the time of study enrollment
* PRIOR THERAPY

  * Patients with recurrent or progressive disease must have received prior chemotherapy, and/or radiotherapy.
  * Patients must have recovered from the acute treatment related toxicities (defined as ≤ Grade 1 if not defined in eligibility criteria; excludes alopecia) prior to entering this study.
  * Patients with newly diagnosed DIPG must have completed radiation therapy
* CHEMOTHERAPY - Patients must have received their last dose of known myelosuppressive anticancer therapy at least 21 days prior to enrollment or at least 42 days if nitrosourea. Patients must have received their last dose of non-myelosuppressive chemotherapy at least 7 days prior to enrollment.
* INVESTIGATIONAL/ BIOLOGIC AGENT:

  * Biologic or investigational agent (anti-neoplastic): Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the investigational or biologic agent ≥ 7 days prior to study enrollment.
  * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
  * Monoclonal antibody treatment and agents with known prolonged half-lives: Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent ≥ 28 days prior to study enrollment.
* RADIATION:

  * Recurrent or Progressive CNS tumor patients must have had their last fraction of:
  * Craniospinal irradiation, whole brain radiation, total body irradiation or radiation to spine ≥ 6 weeks (42 days) prior to enrollment.
  * Focal irradiation ≥ 14 days prior to enrollment.
  * DIPG Patients: Patients with DIPG are eligible after completion of initial radiotherapy (with or without concurrent treatment) and in the absence of progressive disease on post-radiation imaging.
  * Patients must have completed radiation therapy at least 14 days prior to enrollment but no longer than 56 days and cannot have received any other tumor-directed treatment except the following: Patient may have received temozolomide or other non-investigational agents during irradiation at the treating physician's discretion. If the patient has received such agents concurrently with radiation, then patient must have recovered from the acute treatment related toxicities (defined as < Grade 1) prior to enrollment.
* CELLULAR THERAPY: Patient must be:
* ≥ 6 months since allogeneic stem cell transplant prior to enrollment with no evidence of active graft vs. host disease.
* ≥ 3 months since autologous stem cell transplant prior to enrollment.
* > 42 days since completion of any other type of adoptive cellular therapy prior to enrollment.
* CRANIAL SURGERY: Patients who have had recent cranial surgery (VP shunt, ETV, tumor resection) are eligible for inclusion, but the vaccine may not be administered prior to post-operative Day 14.
* NEUROLOGIC STATUS: Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to enrollment. A baseline neurological exam should clearly document the neurological status of the patient at the time of enrollment on the study.
* PERFORMANCE STATUS - Karnofsky Performance Scale (KPS for > 16 years of age) or Lansky Performance Score (LPS for ≤ 16 years of age) assessed within 2 weeks prior to enrollment must be ≥ 60%. Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* ORGAN FUNCTION - Patients must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 0.75 x 109 cells/L
  * Platelets ≥ 100 x 109 cells/L (unsupported, defined as no platelet transfusion within 7 days prior to enrollment)
  * Hemoglobin ≥ 8 g/dl (may receive transfusions)
  * PT/INR, PTT ≤ 1.5 x ULN
  * Total bilirubin ≤ 1.5 times institutional upper limit of normal (ULN)
  * ALT(SGPT) ≤ 3 x institutional upper limit of normal
  * Albumin ≥ 2 g/dl
  * Blood creatinine based on age/gender as noted below. Patients that do not meet the criteria below but have a 24-hour Creatinine Clearance or GFR (radioisotope or iothalamate) ≥ 70 ml/min/1.73 m2 are eligible. Maximum Serum Creatinine for age/gender:
  * Age 1 to < 2 years: 0.6 mg/dL (male); 0.6 mg/dL (female)
  * Age 2 to < 6 years: 0.8 mg/dL (male); 0.8 mg/dL (female)
  * Age 6 to < 10 years: 1 mg/dL (male); 1 mg/dL (female)
  * Age 10 to < 13 years: 1.2 mg/dL (male); 1.2 mg/dL (female)
  * Age 13 to < 16 years: 1.5 mg/dL (male); 1.4 mg/dL (female)
  * Age ≥ 16 years: 1.7 mg/dL (male); 1.4 mg/dL (female)
* INFECTIOUS DISEASES

  * Human Immunodeficiency Virus (HIV) Infected Individuals: Patients who are known to be Human immunodeficiency virus (HIV)-infected must be on effective anti-retroviral therapy with undetectable viral load for 6 months prior to study enrollment.
  * Hepatitis B Chronically Infected Individuals: For patients with known evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
  * Hepatitis C (HCV) Infected Individuals: Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. Patients with known HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load.
* CORTICOSTEROIDS: Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to enrollment. A maximum dose of 0.1 mg/kg/day (and maximum total daily dose 4 mg) of dexamethasone (or equivalent) is permitted at study entry. Effort should be made to reduce to lowest tolerated steroid dose.

Patients must be willing to use brief courses (at least 72 hours) of steroids as directed for potential inflammatory side effects of the therapy if recommended by their treating physician.

* GROWTH FACTORS - Patients must be off all colony-forming growth factor(s) for at least 14 days prior to enrollment (i.e. filgrastim, sargramostim or erythropoietin). Two (2) weeks must have elapsed if the patient received a long-acting formulation.
* PREGNANCY - Pregnant women or nursing mothers are excluded from this study because SurVaxM is an agent with the potential for teratogenic effects. Female patients of childbearing potential must have a negative serum or urine pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* PREGNANCY PREVENTION - Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study.
* INFORMED CONSENT - The patient or parent/guardian is able to understand the consent and is willing to sign a written informed consent document according to institutional guidelines. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

* • BREAST FEEDING WOMEN - Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SurVaxM breastfeeding should be discontinued if the mother is treated with SurVaxM. Female patients who are breastfeeding are not eligible for this study unless they agree not to breastfeed.

Excluded Diagnoses:

* Patients with spinal cord primary tumors
* Patients with relapsed or progressive DIPG
* Patients with metastatic disseminated DIPG are not eligible. MRI of spine must be performed if disseminated disease is suspected by the treating physician.
* Patients with midline high grade gliomas including those with H3 K27M-altered diffuse midline glioma (DMG) centered outside of the pons
* Patients with Grade II myxopapillary ependymoma
* Patients with WHO Grade I or II gliomas are not eligible unless tumor is defined as DIPG as per above.
* Patients with bone-only metastatic lesions that do not have otherwise evaluable CNS disease.

Bulky Disease

Patients with bulky tumor on imaging are ineligible. Bulky tumor is defined as any of the following:

* Tumor with evidence of clinically significant tonsillar herniation
* Tumor with evidence of clinically significant uncal herniation causing midbrain compression or midline shift greater than 5 mm
* Tumor with a diameter >4cm in one dimension on T2/FLAIR
* Tumor that in the opinion of the site investigator, shows significantly rapid progression of mass effect in either the brain or spinal cord such that the priming phase of vaccination (i.e., 6 weeks) cannot be completed before clinical deterioration is likely to occur.

Treating physicians should contact the Study Chair to request a rapid central imaging review to confirm fulfilment of these eligibility criteria, if they have concerns. If clinically appropriate, surgical debulking of large tumors should be considered before study entry.

Concurrent Illness:

* Active, uncontrolled infection requiring treatment (including HIV infection)
* Patients with active autoimmune disease or documented history of autoimmune disease/syndrome that requires ongoing systemic steroids or systemic immunosuppressive agents, with the exception of:
* Patients with vitiligo or resolved asthma/atopy
* Patients with hypothyroidism stable on hormone replacement or Sjogren's syndrome
* History of or ongoing pneumonitis or significant interstitial lung disease
* Patients with any clinically significant unrelated systemic illness (significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results.
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen for this trial.
* Any medical condition that, in the opinion of the Principal Investigator, would compromise the patient's ability to participate in the study.

  • CONCOMITANT MEDICATIONS:
* Patients who are receiving any other anti-cancer or investigational drug therapy are ineligible.
* Patients who are receiving any cannabidiol (CBD) or medical marijuana treatment are ineligible.
* Patients who have received the last vaccination of a live vaccine ≤ 30 days prior to enrollment are ineligible. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and must meet timeline for live vaccine.
* Patients who have received an inactivated virus, peptide, or mRNA vaccine within 14 days of the start of protocol therapy are ineligible.
* Patients may not be on immunosuppressive therapy, including corticosteroids (except as defined in the corticosteroids inclusion criteria) at time of enrollment. However, patients who require intermittent use of bronchodilators, local steroid injections, or topical steroids will not be excluded from the study.
* Patients may not be receiving concomitant chemotherapy, immunotherapy, radiotherapy, radiosurgery, interferon, allergy desensitization injections, growth factors, interleukins, or any investigational therapeutic medication at the time of enrollment.

  * INABILITY TO PARTICIPATE: Patients who in the opinion of the investigator are unwilling or unable to return for required follow-up visits or obtain follow-up studies required to assess toxicity of therapy or to adhere to drug administration plan, other study procedures, and study restrictions.
  * ALLERGY: Known allergy or hypersensitivity to Keyhole Limpet Hemocyanin (KLH), granulocyte colony-macrophage stimulating factor (sargramostim) or MRI contrast agent.
  * BLEEDING DISORDER: Patients with a known coagulopathy or bleeding diathesis or requires the use of systemic, anticoagulant medication are not eligible.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects with Regimen-Limiting Toxicity (RLT) | The first 8 weeks of protocol therapy (6 weeks for 4 priming doses +14 days follow-up from the 4th priming dose)
  The RLT rate during the first 8 weeks (14 days after the 4th priming dose of vaccine) will be used as the primary endpoint for safety monitoring and for determining when enrollment can begin in the next sub-cohort.
Percentage of Subjects with Pseudoprogression Related Regimen-Limiting Toxicity | The first 14 weeks of protocol therapy (6 weeks for 4 priming doses + 8 weeks follow-up from the 4th priming dose)
  A separate RLT assessment window for risk of pseudoprogression will encompass the 6 weeks for administration of 4 priming doses + 8 weeks of follow-up after administration of the 4th priming dose. Pseudoprogression RLTs during this interval will be included in the primary safety monitoring rules and analysis.

SECONDARY OUTCOMES:
Differences in MR permeability and MR perfusion parameters for patients with true progression vs. pseudoprogression | Up to 3 years from treatment initiation.
  Differences in estimated rCBV and ktrans values between patients with pseudoprogression vs. true progression will be reported.

OTHER OUTCOMES:
Best Response Rate | Up to 118 weeks of treatment
  Overall response assessment takes into account response (complete response, partial response, stable disease, progressive disease) in both target and non-target lesion, and the appearance of new lesions, where applicable, according to the criteria described in the protocol. Best radiographic response observed while on treatment will be reported for each patient and percentage of patients that fall in each response category will be reported.
Progression Free Survival | Up to 3 years from treatment initiation
  Interval of time between date of initiation of protocol treatment and minimum date of documentation of Progressive Disease
Overall Survival | Up to 3 years from treatment initiation
  Time between date of initiation of protocol treatment and minimum date of death due to any cause or date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Twist, MD, Study Chair — Roswell Park Comprehensive Cancer Center
Locations (14):
- United States (13):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National, Washington D.C., District of Columbia
  - University of Florida, Gainsville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The Pediatric Brain Tumor Consortium (PBTC) ensures that high dimensional molecular data generated from PBTC samples will be submitted to the NIH Database of Genotypes and Phenotypes (dbGaP) or other NIH-designated data repository. PBTC is required to make data available to other investigators for use in research projects. An investigator requesting data from published PBTC studies will submit a proposal describing the studies from which data are requested, the requested data, and a list of investigators in the project and their affiliated institutions, along with the investigator's CV to the PBTC Steering Committee for review. Once approved, the requesting investigator will be asked to complete a Data Transfer Agreement before the release of deidentified data. Requests for data are typically only considered once the primary study manuscript has been published though exceptions may be made in the event of long delays in the primary study data publication.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 6 months after publication and end timeframe may be up to 10 years.